Ministry of Higher Education and Scientific Research Al-Nahrain University High Institute for Infertility Diagnosis and Assisted Reproductive Technologies





## Study the Effects of Intrauterine flushing with Low Dose Human Chorionic Gonadotrophin on Endometrial Receptivity and ICSI Outcome



OCTOBER 16, 2024

## Consent Form

I, the patient admitted to the Higher Institute for Infertility Diagnosis and Assisted Reproductive Technologies, agree to the intrauterine injection of human chorionic gonadotropin (HCG) by the graduate student Dr. (Omaima Ismail Khalaf) for the purpose of completing her research on the role of intrauterine insemination with human chorionic gonadotropin on the day of egg retrieval in improving the clinical outcomes of IVF patients

Signature